CLINICAL TRIAL: NCT06711874
Title: Clinical Deterioration Caused by Elevated Parathyroid Hormone Levels Among Critically-Ill Patients With Vitamin D Depletion: a Secondary Analysis of a Multicenter, Prospective, Observational Study
Brief Title: Abnormally High Parathyroid Hormone Levels Worsens Outcomes in Vitamin D Depleted Critical Care Patients
Status: Active, not recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202404064RINA
Record Dates: First submitted 2024-11-24; First posted 2024-12-02 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-05

CONDITIONS: Vitamin D Deficiency; Hyperparathyroidism; Critically Ill Patients Admitted in ICU
Keywords: parathyroid hormone; vitamin D depletion; 25(OH)D; critical illness; mortality
MeSH Terms: conditions — Vitamin D Deficiency; Hyperparathyroidism; Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to investigate the impacts of abnormally elevated PTH levels on clinical outcomes among critically ill patients with vitamin D depletion.

DETAILED DESCRIPTION:
This study is a secondary analysis of data from a previous multicentre, prospective, observational cohort study (REC No: 201805087RINB) examining vitamin D deficiency prevalence and outcomes in critical care. From the previously enrolled 651 critically ill patients admitted to medical and surgical intensive care units (ICUs), those enrolled within 48 hours of admission are analyzed. Vitamin D depletion is defined as a serum 25-hydroxyvitamin D (25(OH)D) level <30 ng/mL. Patients are categorized as PTH non-responders (PTH levels of 15-68.3 pg/mL) or PTH responders (PTH levels > 68.3 pg/mL). The primary endpoints include the rate of survival to day 28 and the rate of survival to hospital discharge. Secondary endpoints include the length of ICU stay at day 28 and day 90, Acute Physiology and Chronic Health Evaluation (APACHE) II score, Sequential Organ Failure Assessment (SOFA) score, and blood clinical laboratory variables.

ELIGIBILITY:
Inclusion criteria:

1. Critically ill patients within 48 hours of ICU admission

Exclusion criteria:

1. Less than 20 years old
2. Severe malnutrition (BMI<18kg/m2)
3. Severe anemia (hemoglobin concentration <7g/dL)
4. Receiving high-dose vitamin D treatment (> 3000 IU/day) within four weeks
5. Have been admitted to the ICU within three months
6. Suffering from diseases that affect vitamin D concentration, calcium metabolism or bone metabolism (for example: parathyroid disease, rickets, chirtosis, and severe cirrhosis [Child C])
7. Patients and family members who do not speak the native language

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patient
Sampling Method: Non-Probability Sample
Enrollment: 320 (Estimated)
Dates: Start 2024-05-21 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Mortality | From enrollment to day 90
  Survival on day 28, survival to hospital discharge

SECONDARY OUTCOMES:
Acute Physiology and Chronic Health Evaluation II (APACHE II) score | From enrollment to day 90
  Apache II Score is a severity-of-disease classification system based on a number of laboratory values and patient signs taking both acute and chronic disease into account. An integer score from 0 to 71 with higher scores meaning a worse outcome.
Sequential Organ Failure Assessment (SOFA) score | From enrollment to day 90
  SOFA score is a scoring system that assesses the performance of several organ systems in the body (neurologic, blood, liver, kidney, and blood pressure/hemodynamics) and assigns a score based on the data obtained in each category. An integer score from 0 to 24 with higher scores meaning a worse outcome.
ICU length of stay | From enrollment to day 90
  The days patients stays in ICU
Laboratory parameters | From enrollment to day 90
  Serum levels of 25-hydroxyvitamin D (25(OH)D), calcium, parathyroid hormone (PTH), cortisol

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No